CLINICAL TRIAL: NCT01599663
Title: Pain Management of Intensive Care Unit (ICU) Patients. An Intervention Study to Evaluate the Effect of Systematic Pain Management of Various Groups of ICU Patients.
Brief Title: Pain Management of Intensive Care Unit Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Project number 3234
Record Dates: First submitted 2012-05-04; First posted 2012-05-16 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Pain
Keywords: Pain management; Pain assessment; Intensive care unit; Adult
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention units (Experimental): A time period before the clinicians will be educated, trained and guided in the pain management algorithm, pre-test data will be collected in four ICU units.
  The clinicians in three of the ICU units will be educated, trained and guided in the pain management algorithm. The algorithm will then be used to assess and treat pain in all consecutive ICU patients. Post-test data will be collected a time period after the intervention is implemented.
  Interventions: Other: Pain management algorithm
- Control unit (No Intervention): The clinicians in the fourth ICU (control unit) will not be educated, trained and guided in the pain management algorithm. They will continue to assess and treat pain in all consecutive ICU patients as before. The unit, which will be used as a comparison unit, will collect the same post-test data at the same time as data in intervention ICUs were collected.

INTERVENTIONS:
Other: Pain management algorithm — The algorithm guide the clinicians to score ICU patients pain systematically with different pain assessment tools. The tools are the Numeric Rating Scale, Behavioral Pain Scale and Behavioral Pain Scale Non Intubated. The algorithm guide the clinicians to choose between the different pain assessment tools depending on the ICU patient's condition and ability to rate his own pain. Thereafter the algorithm guide the clinicians to treat pain depending on the pain intensity score.
  Arms: Intervention units

SUMMARY:
The purpose of this study is to evaluate the effect of an algorithm, where ICU patients pain are assessed systematically with valid pain assessment tools and where pain is treated after pain intensity score.

DETAILED DESCRIPTION:
As a pre-test, before the intervention is introduced, data from ICU patients from four intensive care units (ICU) will be collected from medical records to evaluate current pain management practices. An algorithm, which is developed by a group of resource persons, is educated to the staff in three of the ICUs. The staff will also receive training and guiding in the use of the algorithm and the different pain assessment tools. Then the algorithm will be implemented and used in all the consecutive ICU patients. Post-test data is then collected in the three ICUs. In the fourth ICU, which will be used as a comparison unit, the same post-test data will be collected at the same time as data in intervention ICUs were collected. The algorithm will not be introduced here.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients admitted into these four ICUs

Exclusion Criteria:

* Patients will be excluded if they are not able to express pain behaviors (i.e. quadriplegic, are receiving neuromuscular blockade or muscle paralyzing drugs or are being investigated for brain death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2012-05; Primary Completion 2017-05 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation, ICU and hospital length of stay | The participants will be followed for the duration of hospital stay, an expected average of two weeks
  Duration of mechanical ventilation, ICU and hospital length of stay will be measured in a group of ICU patients before (pre-test) and after (post-test) the intervention.

SECONDARY OUTCOMES:
Documentation of ICU patients' pain and pain management in four ICU's. | The participants will be followed for the duration of ICU stay, an expected average of one week
  The data is collected to evaluate current pain and pain management practices in a period before the intervention is implemented (pre-test). The data is collected from both intervention units and control unit.
Proportion of ICU patients express having pain or are estimated to have pain. How severe their pain is. | The participants will be followed for the duration of ICU stay, an expected average of one week
  In the pre-test, the medical records are searched for use of different pain assessment tools or other notations about pain assessment of these patients. In the post-test the medical records are searched for systematically pain intensity scores from the different pain assessment tools.
The clinician's adherence to the pain management algorithm in ICU patients. | The adherence will be followed for the duration of ICU stay, an expected average of one week (post-test)
  The medical records will be searched for documentation of how the algorithm is used. I.e. is it used to the right patients, Is it used as often as described, is it used to the right patients.
Sedation level and Use of psychoactive drugs | The participants will be followed for the duration of ICU stay, an expected average of one week
  Sedation level and use of psychoactive drugs will be measured before (pre-test) and after (post-test) the intervention.
Use of Analgesics | The participants will be followed for the duration of ICU stay, an expected average of one week
  Use of analgesics will be measured before (pre-test) and after (post-test) the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Brita F Olsen, Msc, Principal Investigator — Ostfold Hospital Trust
Locations (1):
- Ostfold Hospital Trust, Fredrikstad, Norway

IPD SHARING:
Plan to Share IPD: No